CLINICAL TRIAL: NCT01396655
Title: Analysis of Clinical Outcome, Predictive and Prognostic Factors of Therapeutic Responses in Patients Who Treated With Doxorubicin & Docetaxel Neoadjuvant Chemotherapy in Clinical Stage II or III Breast Cancer
Brief Title: PET in Breast Cancer Receiving Neoadjuvant Chemotherapy
Acronym: DA-PET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seock-Ah Im, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA-PET-2010-0022299
Record Dates: First submitted 2011-06-16; First posted 2011-07-19 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2011-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant chemotherapy; molecular marker; FDG PET; locally advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- docetaxel + doxorubicin (Experimental): The chemotherapeutic regimen consisted of docetaxel (75 mg/m2) and doxorubicin (50 mg/m2) by intravenous infusion every 3 weeks.
  Interventions: Drug: docetaxel (75 mg/m2) and doxorubicin (50 mg/m2)

INTERVENTIONS:
Drug: docetaxel (75 mg/m2) and doxorubicin (50 mg/m2) — The chemotherapeutic regimen consisted of docetaxel (75 mg/m2) and doxorubicin (50 mg/m2) by intravenous infusion every 3 weeks. After three cycles of neoadjuvant chemotherapy, the patients were re-evaluated for response and underwent curative surgery. Radiologic response was evaluated using breast magnetic resonance imaging (MRI) for the primary breast tumor and chest computed tomography (CT) for axillary, supraclavicular, internal mammary lymph nodes with RECIST criteria. Both breast MRI and chest CT were performed in all the 78 patients. Subsequently, the patients received three more cycles of docetaxel and doxorubicin as an adjuvant chemotherapy, followed by hormonal or radiation therapy, if indicated.

SUMMARY:
Prognostic factors in locally advanced breast cancer treated with neoadjuvant chemotherapy differ from those of early breast cancer.

The purpose of this study was to identify the clinical significance of potential predictive and prognostic factors including serial FDG PET/CT in breast cancer patients treated by neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically-confirmed breast cancer by core needle biopsy,
2. initial clinical stage II or III,
3. objective measurable lesion,
4. ECOG performance 0~2,
5. previously untreated,
6. adequate bone marrow, hepatic, cardiac, and renal functions
7. age 20~70
8. agreement with this trial, and written informed consent

Exclusion Criteria:

1. history of other cancer
2. active infection
3. pregnancy
4. psychologic disease
5. uncontrolled heart diseases
6. male

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
pathologic complete response | after completion of 3 cycles of neoadjuvant chemotherapy (9 weeks after initiation of chemotherapy)
  The primary end point of this trial was evaluating pathologic complete response (pCR) rate. After 3 cycles of neoadjuvant chemotherapy, patients were undertook breast surgery. Using post operative pathology specimen, we evaluated pathologic response and calculated pCR rate.

SECONDARY OUTCOMES:
survival (Relapse-free survival, overall survival) | 2years , 3 years and 5 years after initiation of neoadjuvant chemotherapy
  Relapse-free survival, overall survival were estimated by Kaplan-Meier product limit methods
early metabolic response | before chemotherapy, and after 1cycle of neoadjuvant chemotherapy (15th days after 1cycle)
  Early metabolic response were evaluated by serial FDG PET/CT before and after 1cycle of neoadjuvant chemotherapy (15th days after 1cycle). Declining of SUV were calculated
predictive factors | after completion of 3 cycles of neoadjuvant chemotherapy (9 weeks after initiation of chemotherapy)
  Predictive factors for pathologic complete response were analyzed using univariate and multivariate logistic regression analysis
hematologic toxicity | every q 3weeks during chemotherapy (up to 24 weeks from initiation of chemotherapy)
  Hematologic toxicities are evaluated every q 3weeks during chemotherapy. Neutropenia,thrombocytopenia, and anemia are evaluated during chemotherapy (per cycles) by NCI CTCAE v3.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bhumsuk Keam, MD, Principal Investigator — Seoul National University Hospital; Seock-Ah Im, MD PhD, Principal Investigator — Seoul National University Hospital

REFERENCES:
- [Derived] Keam B, Im SA, Koh Y, Han SW, Oh DY, Cho N, Kim JH, Han W, Kang KW, Moon WK, Kim TY, Park IA, Noh DY, Chung JK, Bang YJ. Early metabolic response using FDG PET/CT and molecular phenotypes of breast cancer treated with neoadjuvant chemotherapy. BMC Cancer. 2011 Oct 20;11:452. doi: 10.1186/1471-2407-11-452. PMID 22011459